CLINICAL TRIAL: NCT01183858
Title: A Prospective, Double-blind Randomized Phase III Study of 300 mg Versus 150 mg Erlotinib in Current Smokers With Locally Advanced or Metastatic NSCLC in Second-line Setting After Failure on Chemotherapy (CURRENTS)
Brief Title: A Study of Tarceva (Erlotinib) to Compare Two Different Doses in in Currently Smoking Patients With Advanced or Metastatic Non-Small Cell Lung Cancer (CURRENTS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MO22162; 2010-018476-24 (EudraCT Number)
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Erlotinib 150 mg (Experimental): Erlotinib 150 mg single daily oral dose until disease progression.
  Interventions: Drug: Erlotinib [Tarceva]
- Erlotinib 300 mg (Experimental): Erlotinib 300 mg single daily oral dose until disease progression.
  Interventions: Drug: Erlotinib [Tarceva]

INTERVENTIONS:
Drug: Erlotinib [Tarceva] — Single daily oral dose
  Other Names: Tarceva

SUMMARY:
This prospective, double-blind, randomized study will evaluate the safety and efficacy of two dose levels of erlotinib [Tarceva] on progression-free survival, response and disease control rates and overall survival in patients with advanced or metastatic non-small cell lung cancer (NSCLC) after failure of first-line platinum-based chemotherapy. Patients must be current smokers and not intending to stop smoking during the study. Patients will be randomized to receive either 150 mg or 300 mg of study drug as single daily oral doses. Treatment will continue until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years
* inoperable, locally advanced (stage IIIB/IV) with supraclavicular lymph node metastases or malignant pleural or pericardial effusion) or metastatic (stage IV) non-small cell lung cancer (NSCLC)
* Disease must be characterized according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Patients have received one prior platinum-based chemotherapy regimen for advanced NSCLC, but must have recovered from any treatment-related toxicity
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥12 weeks
* Current cigarette smoker (having smoked >100 cigarettes in entire lifetime and currently smoking on average ≥1 cigarette per day), not intending to stop during the study

Exclusion Criteria:

* Prior antibody or small molecule therapy against Epidermal growth factor receptor (EGFR)
* Radiotherapy within 28 days prior to enrollment
* Received more than one line of chemotherapy for locally advanced/metastatic NSCLC (first-line maintenance chemotherapy after first-line platinum-based chemotherapy is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (53):
- China (11):
  - Beijing
  - Changchun
  - Chengdu
  - Fuzhou
  - Guangzhou
  - Nanjing
  - Nanning
  - Shanghai
  - Shenyang
  - Tianjin
  - Wuhan
- Denmark (4):
  - Copenhagen
  - Hillerød
  - Næstved
  - Roskilde
- Cairo, Egypt
- France (5):
  - Caen
  - Limoges
  - Marseille
  - Paris
  - Pontoise
- Germany (13):
  - Berlin
  - Essen
  - Gauting
  - Großhansdorf
  - Hanover
  - Immenhausen
  - Lostau
  - München
  - Nuremberg
  - Rheine
  - Villingen-Schwenningen
  - Wuppertal
  - Würselen
- Netherlands (4):
  - Amsterdam
  - Breda
  - Nieuwegein
  - Zwolle
- Spain (6):
  - Barcelona, Barcelona
  - Sabadell, Barcelona, Barcelona
  - Madrid, Madrid
  - Málaga, Malaga
  - Seville, Sevilla
  - Valencia, Valencia
- Switzerland (4):
  - Baden
  - Basel
  - Bern
  - Fribourg
- Turkey (Türkiye) (5):
  - Ankara
  - Eskişehir
  - Gaziantep
  - Izmir
  - Konya

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 315 participants were randomized. 313 participants were included in the Intent-to -treat (ITT) population. The ITT population excluded 2 randomized participants: 1 participant randomized in error and 1 participant with missing source data.
Period: Overall Study
Arm/Group | Erlotinib 150 mg | Erlotinib 300 mg
Started | 154 | 159
Safety Population | 154 | 158
Completed | 1 | 3
Not Completed | 153 | 156
Not completed — Death not related to Progressive Disease | 5 | 6
Not completed — Adverse Event | 14 | 11
Not completed — Investigator's Decision | 0 | 3
Not completed — Insufficient Therapeutic Response | 2 | 0
Not completed — Refused Treatment | 1 | 4
Not completed — Withdrew Consent | 4 | 4
Not completed — Discontinued Smoking | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Administrative/Other | 6 | 6
Not completed — Progressive Disease | 112 | 115
Not completed — Death related to Progressive Disease | 4 | 5
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat Population included all randomized participants. 2 participants were excluded from analysis: 1 participant randomized in error and 1 participant with missing source data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib 150 mg | Erlotinib 300 mg | Total
Number analyzed (Participants) | 154 | 159 | 313
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (9.25) | 59.2 (9.14) | 59.4 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 120 | 124 | 244

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the date of first occurrence of disease progression or death. For target lesions, Progressive Disease (PD) was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Randomization to Clinical Cutoff: 28 October 2013 (Up to 36.5 Months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib 150 mg | Erlotinib 300 mg
Number analyzed (Participants) | 154 | 159
weeks | 6.86 [6.29 to 12.00] | 7.00 [6.29 to 11.00]
Statistical Analysis 1: Comparison: Erlotinib 150 mg vs Erlotinib 300 mg; Test type: Superiority or Other; p = 0.671, Log Rank — Unstratified analysis; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.83 to 1.33]

2. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from randomization to the date of death due to any cause.
Time Frame: Randomization to Clinical Cutoff: 28 October 2013 (Up to 36.5 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib 150 mg | Erlotinib 300 mg
Number analyzed (Participants) | 154 | 159
months | 6.77 [5.65 to 8.77] | 6.83 [5.39 to 8.48]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Tumor response was assessed by the investigator using computer tomography (CT) or magnetic resonance imaging (MRI) scans according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. A participant was defined as a responder if they sustained a complete response (CR) or partial response (PR) for at least 4 weeks during randomized treatment (confirmed response). Patients with no tumor assessment after the start of study treatment were to be considered as non-responders. The percentage of participants in each best response category is presented.
Time Frame: Randomization to Clinical Cutoff: 28 October 2013 (Up to 36.5 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib 150 mg | Erlotinib 300 mg
Number analyzed (Participants) | 154 | 159
percentage of participants
  Complete Response | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Partial Response | 7.1 [3.6 to 12.4] | 2.5 [0.7 to 6.3]
  Stable Disease | 33.1 [25.8 to 41.1] | 34.0 [26.6 to 41.9]
  Progressive Disease | 44.8 [36.8 to 53.0] | 45.9 [38.0 to 54.0]
  Not Evaluable | 14.9 [9.7 to 21.6] | 17.6 [12.0 to 24.4]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Tumor response was assessed by the investigator using computer tomography (CT) or magnetic resonance imaging (MRI) scans. Disease control rates were measured according to RECIST version 1.1 criteria. A participant was defined as having controlled disease if they sustained a Complete Response (CR) or Partial Response (PR) for at least 4 weeks during randomized treatment (confirmed response), or Stable Disease (SD) for at least 6 weeks. Patients with no tumor assessment after the start of study treatment were considered as having uncontrolled disease. The percentage of participants with Disease Control is presented.
Time Frame: Randomization to Clinical Cutoff: 28 October 2013 (Up to 36.5 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib 150 mg | Erlotinib 300 mg
Number analyzed (Participants) | 154 | 159
percentage of participants | 40.3 [32.4 to 48.5] | 36.5 [29.0 to 44.5]

5. Secondary Outcome: Time to Progression (TTP)
Description: Tumor response was assessed by the investigator using computer tomography (CT) or magnetic resonance imaging (MRI) scans according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria. Time to progression (TTP) in weeks was defined as the time from randomization to the date of disease progression. Participants without event were censored at the date of the last tumor assessment when the patient was known to be progression free.
Time Frame: Randomization to Clinical Cutoff: 28 October 2013 (Up to 36.5 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib 150 mg | Erlotinib 300 mg
Number analyzed (Participants) | 154 | 159
weeks | 9.86 [6.43 to 12.14] | 9.14 [6.43 to 12.00]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) at the End of the Study
Description: An adverse event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events.
  A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
  Adverse Events in the following categories are presented: Adverse Events, Serious Adverse Events, AEs leading to withdrawal from treatment and AEs leading to death.
Time Frame: Randomization to End of Study: 14 October 2010 - 7 February 2014 (Up to 39.8 months)
Population: Safety population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Erlotinib 150 mg | Erlotinib 300 mg
Number analyzed (Participants) | 154 | 158
participants
  Adverse Events (AEs) | 130 | 141
  Serious Adverse Events | 29 | 35
  AEs leading to withdrawal | 18 | 15
  AEs leading to death | 12 | 13

7. Primary Outcome: Progression-Free Survival (PFS) at the End of Study
Description: as for outcome 1
Time Frame: Randomization to End of Study: 14 October 2010 - 7 February 2014 (Up to 39.8 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib 150 mg | Erlotinib 300 mg
Number analyzed (Participants) | 154 | 159
weeks | 6.86 [6.29 to 12.00] | 7.00 [6.29 to 11.43]
Statistical Analysis 1: Comparison: Erlotinib 150 mg vs Erlotinib 300 mg; Test type: Superiority or Other; p = 0.625, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.84 to 1.33]

8. Secondary Outcome: Overall Survival (OS) at the End of Study
Description: OS defined as the time from randomization to the date of death due to any cause.
Time Frame: Randomization to End of Study: 14 October 2010 - 7 February 2014 (Up to 39.8 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib 150 mg | Erlotinib 300 mg
Number analyzed (Participants) | 154 | 159
months | 7.00 [5.65 to 8.84] | 6.90 [5.62 to 8.64]

ADVERSE EVENTS:
Time Frame: Randomization to End of Study: 14 October 2010 - 7 February 2014 (Up to 39.8 months)
Description: Safety population: All participants who received at least 1 dose of study drug.
Arm/Group | Erlotinib 150 mg | Erlotinib 300 mg
Serious Adverse Events (participants affected / at risk) | 29/154 | 35/158
Other Adverse Events (participants affected / at risk) | 115/154 | 128/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib 150 mg (N=154) | Erlotinib 300 mg (N=158)
Pneumonia (Infections and infestations) | 6 | 3
Respiratory tract infection (Infections and infestations) | 0 | 3
Anal abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 3
Fatigue (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 3
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib 150 mg (N=154) | Erlotinib 300 mg (N=158)
Rash (Skin and subcutaneous tissue disorders) | 43 | 75
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 16
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 11 | 9
Diarrhoea (Gastrointestinal disorders) | 29 | 46
Nausea (Gastrointestinal disorders) | 20 | 17
Vomiting (Gastrointestinal disorders) | 13 | 14
Constipation (Gastrointestinal disorders) | 9 | 11
Dyspepsia (Gastrointestinal disorders) | 3 | 8
Abdominal pain upper (Gastrointestinal disorders) | 1 | 8
Fatigue (General disorders) | 21 | 26
Chest pain (General disorders) | 7 | 14
Asthenia (General disorders) | 9 | 12
Pain (General disorders) | 8 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 19
Decreased appetite (Metabolism and nutrition disorders) | 26 | 32
Weight decreased (Investigations) | 7 | 15
Anaemia (Blood and lymphatic system disorders) | 6 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 8
Headache (Nervous system disorders) | 9 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.